CLINICAL TRIAL: NCT06773637
Title: Introduction of a Standardized Novel Periapical Radiography Technique for Long Term Follow up of Implants Inserted Simultaneously With Sinus Allogenic Bone Augmentation: A Retrospective Study of a Case Series.
Brief Title: A Standardized Novel Periapical Radiography Technique for Long Term Follow up of Implants Inserted Simultaneously With Sinus Allogenic Bone Augmentation
Status: Completed | Type: Observational
Sponsor: Misr International University (Other)
Collaborators: Suez Canal University (Other)
Responsible Party: Principal Investigator, Hebatallah Abdo's Elsaid Mattar, Assistant Lecturer Oral & Maxillofacial Surgery Department, Misr International University
Other Study IDs: 2024/842
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Open Sinus Elevation; Periapical Radiograph
Keywords: periapical radiograph; dental implants; open sinus elevation; closed sinus elevation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Aim of this study is introducing a standardized novel periapical radiography technique for long term follow up of implants inserted simultaneously with sinus allogenic bone augmentation.

This novel standardized periapical radiographic technique was introduced and has been performed on patients who were already enrolled in a study performed at Suez Canal University. This aforementioned study was conducted in fulfillment of a PHD thesis that had the ethical approval number of 419/2021.

In that study according to its sample size calculation, 30 implants were tested for a long term, 1 year follow up after having undergone open or closed sinus elevation as a surgical procedure (according to the random sequence generated at that time). In addition to simultaneous implant placement and allogenic bone grafting. Hence for the purpose of accurate measurement of mesial and distal marginal bone changes for these implants over the different follow up intervals and up to one year after implant placement a standardized jig had to be created. This jig had to be customized for each patient and had to maintain its shape and integrity and patient position every time a periapical radiograph was performed. These patients were followed up using this radiographic technique immediate postoperatively, 3, 9 and 12 months postoperatively to evaluate the mesial and distal marginal bone levels according to the previously mentioned study protocol.

DETAILED DESCRIPTION:
Introduction and Review of literature The success of dental implants had been for so long identified by variable criteria. (1). However radiographic measurement of marginal bone levels and its loss had always been consistently one of them (2). Intraoral standardized periapical radiography was always the method of choice for such measurement (3).

Paralleling technique is the foundation of an ideal periapical radiograph, since errors in determining the marginal bone height result from any deviation from the proper vertical angle. The use of an aiming and stabilizing device for the film with a silicone bite registration can be very useful for subsequent measurements and comparisons of marginal bone losses (4). However, it has been noted that the visual interpretation of intraoral radiographs has limited diagnostic relevance for the early detection of small changes in bone. That is due to the fact that before alterations in conventional radiographs become visible, roughly 30 to 50% of bone mineral must be lost (5).

Therefore, various techniques for evaluating alveolar bone height have been widely applied in periodontal and implant research. Direct measurements using graded rulers with millimeters or more complex techniques using computer software and digital imagery had been used widely in the literature. While the digital softwares available for evaluation of marginal bone levels have been proven to be very efficient and accurate to use (6).

The use of the DIGORA for Windows (DFW) software was proposed in the literature frequently associated with accurate measurements of marginal bone levels around dental implants. As well as for its significance of density measurements. (7). For many years now, digital radiography has been proved as an accurate tool in detecting small changes in bone density. Consequently, it was found to be suitable for assessing bone healing (8).

It offers several advantages over conventional films mainly is that digital radiographs offer 80 % reduction in radiation doses, time saving, the elimination of dark room procedures, real-time image display, and opportunities for tele-consultations with radiologists are well known to be cost-effective and reliable. The main advantage of digital techniques that is not shared by conventional radiography is that images are not static, but may be, manipulated by image processing to enhance diagnosis (9).

In the studies of maxillary sinus floor elevation with dental implants placement the use of digitally performed standardized periapical radiographs to measure the marginal bone levels gain or loss had been documented in the literature (10).

And in these studies, and other studies using the modality of intra-oral standardized radiography for assessment of marginal bone levels around placed dental implants, the accepted protocol for measurements follow up was usually based on a 3-month analysis such as immediately postoperative, 3 months and 6 months. (11).

Aim of the study The Aim of this study is introducing a standardized novel periapical radiography technique for long term follow up of implants inserted simultaneously with sinus allogenic bone augmentation.

Materials and Methods

Study Population:

This novel standardized periapical radiographic technique was introduced and has been performed on patients who were already enrolled in a study performed at Suez Canal University. This aforementioned study was conducted in fulfillment of a PHD thesis that had the ethical approval number of 419/2021.

In that study according to its sample size calculation, 30 implants were tested for a long term, 1 year follow up after having undergone open or closed sinus elevation as a surgical procedure (according to the random sequence generated at that time). In addition to simultaneous implant placement and allogenic bone grafting. Hence for the purpose of accurate measurement of mesial and distal marginal bone changes for these implants over the different follow up intervals and up to one year after implant placement a standardized jig had to be created. This jig had to be customized for each patient and had to maintain its shape and integrity and patient position every time a periapical radiograph was performed. These patients were followed up using this radiographic technique immediate postoperatively, 3, 9 and 12 months postoperatively to evaluate the mesial and distal marginal bone levels according to the previously mentioned study protocol.

Preparation of the radiographic bite jig for standardized periapical radiographs Mesial and distal marginal bone levels were measured using a standardized periapical software using the the KaVo Scan eXam OneTM intraoral digital imaging photostimulable phosphor (PSP) plate system which is a film-like thin, flexible, and wireless phosphorescent plate and works as a wireless receptor. This plate will be held by a paralleling device suitable to act as a film holder for it which is the extension cone paralleling (XCP) device namely the Rinn XCP-PSP Fit® to facilitate long cone paralleling techniques. However, to standardize the images measurements a radiographic occlusal bite jig was constructed preoperatively and saved for all following visits in accordance with those constructed in the literature for this purpose (12,13).

However, we used in our study rubber base impression material namely ZetaplusTM (condensation silicone elastomeric material) instead of the wax proposed by (12) to ensure its stability for all the following follow up visits.

Outcomes assessment:

Mesial and Distal Marginal bone level:

Marginal bone level was measured at T1, T2, T3 and T4 follow up periods, by using a standardized periapical radiograph using paralleling device film holders and a customized occlusal jig to hold a PSP digital x ray film as was explained before.

The mesial and distal marginal bone levels were recorded at each of the follow up periods by measuring the length on the CLINIVIEWTM software between the implant platform and the highest visible bone level at the mesial and distal levels of the implant.

Statistical analysis

Experimental design and data analysis:

All collected data will be calculated, tabulated, and statistically analyzed using suitable statistical tests as follows.

1. A normality test will be done to check normal distribution for data by Shapiro-Wilk test.
2. Descriptive statistics will be calculated in the form of Mean ± Standard deviation (SD), range (Max- Min). Qualitative data will be presented as frequencies (n) and percentages (%).
3. ANOVA - test or Kruskal-Wallis test (According to the types of data) One-way ANOVA (Analysis of variance) will be used to compare between time interval (more than two intervals). Tukey post-hoc test or other post hoc tests will be performed for the evaluation of statistical significances among the groups.
4. T- test or Mann-Whitney test (According to the types of data) Independent Student's T-test or Mann-Whitney will be performed for the mean differences between the two groups for normally distributed and not normally distributed respectively.
5. P<0.05 is considered significant.
6. Statistical analysis will be performed using the computer program SPSS software for windows version 26.0 (Statistical Package for Social Science, Armonk, NY: IBM Corp)

ELIGIBILITY:
Inclusion Criteria:

* 1. Males and females ≥ 18 years of age. 2. ASA I and ASA II. 3. Patients having partial edentulism in the posterior region of the maxilla. 4. Edentulous sites consist of native non augmented bone. 5. Horizontal ridge dimension minimum of 5mm 6. The vertical ridge dimension 4-7 mm. 7. Bone quality of D2 or D3. 8. Enough inter-arch distance. 9. The presence of one-year postoperative radiograph CBCT. 10. Presence of postoperative follow up clinical data.

Exclusion Criteria:

* 1. Patients with active acute infection or residual lesion related to the edentulous sites. 2. Acute maxillary sinus pathosis 3. A remaining root dislodged in the Maxillary sinus. 4. Patients that lack a stable occlusion or have parafunctional habits. 5. Patients with poor oral hygiene who are not amenable to motivation and improvement. 6. Smokers who smoke more than 10 cigarettes a day. 7. Pregnant or lactating mothers. 8. Alcohol and drug abuse. 9. Treatment with radiation therapy in the craniofacial region within the previous 12 months

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This novel standardized periapical radiographic technique was introduced and has been performed on patients who were already enrolled in a study performed at Suez Canal University. This aforementioned study was conducted in fulfillment of a PHD thesis that had the ethical approval number of 419/2021.
  In that study according to its sample size calculation, 30 implants were tested for a long term, 1 year follow up after having undergone open or closed sinus elevation as a surgical procedure (according to the random sequence generated at that time). In addition to simultaneous implant placement and allogenic bone grafting. Hence for the purpose of accurate measurement of mesial and distal marginal bone changes for these implants over the different follow up intervals and up to one year after implant placement a standardized jig had to be created. This jig had to be customized for each patient and had to maintain its shape and integrity and patient position every time a periapical
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Mesial and Distal Marginal bone level: | 1 year
  Marginal bone level was measured at T1, T2, T3 and T4 follow up periods, by using a standardized periapical radiograph using paralleling device film holders and a customized occlusal jig to hold a PSP digital x ray film as was explained before.
  The mesial and distal marginal bone levels were recorded at each of the follow up periods by measuring the length on the CLINIVIEWTM software between the implant platform and the highest visible bone level at the mesial and distal levels of the implant.

CONTACTS AND LOCATIONS:
Locations (1):
- Oral & Maxillofacial Surgery Department, Faculty of Dentistry, Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided